CLINICAL TRIAL: NCT06538987
Title: Anesthetic Management in Patients Undergoing Epicardial Ablation for the Treatment of Ventricular Tachycardia; Retrospective Study
Brief Title: Anesthetic Management in Patients Undergoing Epicardial Ablation
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ferda YAMAN, Associate Professor, Eskisehir Osmangazi University
Other Study IDs: EskisehirU
Record Dates: First submitted 2024-07-08; First posted 2024-08-06 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-03

CONDITIONS: Ventricular Tachycardia
Keywords: anesthesia; ventricular tachycardia; Electrophysiology; electro-anatomic mapping; catheter ablation; risk assessment
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: percutaneous epicardial ablation — Epicardial catheter ablation is often necessary for the successful treatment of scar-induced ventricular tachycardia (VT), especially in patients with nonischemic cardiomyopathy (NICMP) where scarring is more extensive on the mid-myocardial or epicardial surface. Because epicardial mapping can be painful and patient movement can limit mapping and safe epicardial access, a common strategy for these patients is general anesthesia.

SUMMARY:
The study is a retrospective study and is descriptive in nature. In this study, the investigators aimed to emphasize the importance of anesthesia management by cardiac risk assessment of patients undergoing epicardial ablation under general anesthesia and analysis of complications that developed during the procedure.

DETAILED DESCRIPTION:
The study is retrospective observational and data were collected by examining the files of all epicardial ablation patients received in the angiography unit starting from 30.10.2020 until 30.10.2022 after ethics committee approval is obtained. Baseline characteristic features of the patients Sex, Age, (years, BMI (kg/m2) Hypertension, Coronary artery disease, COPD (Chronic obstructive pulmonary disease), CKD (Chronic kidney disease) Electrical storm, and ventricular tachycardia etiology, Ischemic cardiomyopathy, Dilated cardiomyopathy, the presence of ARVC (Arrhythmogenic Right Ventricular Cardiomyopathy), Hypertrophic cardiomyopathy will be recorded. NHYA classification will be examined in two groups as NHYA I or II and NHYA III or IV, also estimated glomerular filtration rate, left ventricular ejection fraction, PAAINESD (acute hemodynamic decompensation risk assessment score), iVT score (Risk of VT recurrence) Score information will be recorded. Ventricular tachycardia focus locations, dopamine, dobutamine, norepinephrine infusion requirement during the procedure, arrest development during the procedure, fluoroscopy time and ablation times will be recorded. In the follow-up of the patients after the procedure Causes of death, decompensated heart failure, transient ischemic attack, development of acute renal failure, and recurrence of ventricular tachycardia will be recorded. PAAINESD score (acute hemodynamic decompensation risk assessment score) will be recorded. The PAAINESD Score, developed to estimate the risk of periprocedural hemodynamic decompensation, has values ranging from 0 to 35 points (or 0 to 31 [PAINESD] when the modifiable intraprocedural variable "general anesthesia" is excluded). duration of the procedure, the need for inotropes during the procedure, whether the patient needed mechanical ventilation after the procedure, and the success rates after the procedure will be recorded.

PAINESD Pulmonary disease (chronic obstructive pulmonary disease) 5 Age >60 years 3 Anaesthesia (general) 4 Ischaemic cardiomyopathy 6 NYHA class III or IV 6 Ejection fraction <25 % 3 Storm (VT). 5 Diabetes 3 Data will be analyzed in three separate categories, the characteristics of the patients before the procedure, during the procedure and after the procedure. Descriptive tables and percentages of parameters will be created by statistical analysis.

ELIGIBILITY:
Inclusion Criteria: • age > 18 years old who underwent elective VT ablation between 2020 - 2022,

* primary anesthetic type listed as general anesthesia

Exclusion Criteria: • age < 18 years,

* missing follow-up data,
* patients who have previously undergone epicardial ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Since it is a retrospective study, patients who underwent epicardial ablation within the specified date range will be included. Although the estimated number of cases cannot be predicted, it is a rare and specialized procedure. No group has been determined, the characteristics of the patients and their anesthesia management will be examined in an observational study.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
sex | 2 years
  male %
age | 2 years
  years
weight | 2 years
  kilograms
height | 2 years
  meters
Hypertension | 2 years
  yes or no
Diabetes mellitus | 2 years
  yes or no
Coronary artery disease | 2 years
  yes or no
Chronic obstructive pulmonary disease | 2 years
  yes or no
Chronic kidney disease | 2 years
  yes or no
Systolic pulmonary artery pressure | 2 years
  mmHg
Left ventricular ejection | 2 years
  %
PAAINESD (Acute hemodynamic decompensation risk assessment, ranging from 0 to 35 points, 35 point is the worst) score | 2 years
  score 0-35
ASA ( American Society of Anesthesiologists (ASA) physical status classification ranging from I to IV | 2 years
  score I-IV
Hemoglobin | 2 years
  g/dl
glomerular filtration rate (eGFR) | 2 years
  ml/dak/1,73m2
Total procedural time | 2 years
  minutes
Fluoroscopy time | 2 years
  minutes
Ablation time | 2 years
  minutes

SECONDARY OUTCOMES:
Transient ischemic attack after procedure | 2 years
  yes or no
Exitus during the follow-up | 2 years
  yes or no
cause of death | 2 years
  End-Stage heart failure, VT storm

CONTACTS AND LOCATIONS:
Overall Officials: ferda yaman, Assoc prof, Principal Investigator — University of Eskişehir Osmangazi
Locations (1):
- University of Eskisehir Osmangazi, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided